CLINICAL TRIAL: NCT00951678
Title: Determination of Anatomic Variations of the Internal Jugular and Femoral Veins Using Ultrasound in the Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tampa General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 106983
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Vascular Anatomy
Keywords: ultrasound; femoral vein; internal jugular vein

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ER patients: Subjects must be 18 yrs or older, male or female, and must have the anatomy that we will be examining. Patients will be given the option of enrolling in the study whilst being cared for in Tampa General Hospital Emergency Room.
  We anticipate enrolling normal, healthy volunteers, elderly persons (>65) not cognitively impaired, persons with social, economic or educational disadvantages , and persons who do not understand English fluently.
  Interventions: Other: Observational ultrasonography of venous anatomy

INTERVENTIONS:
Other: Observational ultrasonography of venous anatomy — The patient will have ultrasound images obtained of the right and left internal jugular veins as a function of the degree of head rotation and of the right and left femoral veins. Our study is an observational study

SUMMARY:
Central venous catheterization is a common and important procedure done in the emergency department. The internal jugular vein (IJV), subclavian vein (SV) and femoral vein (FV) are commonly used for central venous access. Unfortunately, this procedure has high-risk complications.

Traditionally, physicians have relied on the use of anatomic landmarks and physical manipulation such as moving the head or rotating the leg in order to place central catheters; however, studies have demonstrated that significant anatomic variations exist within large percentages of study populations. In addition, although studies have demonstrated that the use of ultrasonography for placement of femoral catheters leads to lower rates of complications, no previous studies have specifically determined anatomic variations in the femoral triangle. Therefore, this study will examine the anatomic variation of the IJV vs. carotid artery and the femoral vein vs. femoral artery in the emergency room setting. The investigators will study the variation as a function of sex, age, race, body habitus and degree of head rotation (measured using a goniometer) and in doing so, the investigators will demonstrate the utility of using ultrasound to place central lines in order to decrease morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Patients being cared for in the Tampa General Hospital Emergency Department
* 18 yrs or older
* male or female
* have the anatomy that will be examined (lateral neck and femoral regions)
* speak either English or Spanish
* alert and oriented to person, place, time and situation
* stable vital signs

Exclusion Criteria:

* under 18 yrs
* incarcerated individuals
* those with acute changes in mental status (intoxicated, encephalopathy, psychosis)
* those from whom consent could not be obtained
* those requiring intensive care monitoring
* persons having pathologies that would interfere with the ultrasound investigation
* persons who do not speak English or Spanish
* persons with acute or severe mental or cognitive disabilities
* individuals in a sedated, traumatized or crisis state

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Emergency room patients who fit inclusion criteria and consent to participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
To determine the variability that exists within the vascular anatomy of the lateral neck and femoral regions | Within the timeframe of the study

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Derr, MD, Principal Investigator — USF Emergency Medicine Residency Program
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States